CLINICAL TRIAL: NCT02571244
Title: Telephone Counseling and Text Messaging for Supporting Post-discharge Quit Attempts Among Hospitalized Smokers in Brazil
Brief Title: Text Messaging for Supporting Quit Attempts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Juiz de Fora (Other)
Collaborators: University of Kansas (Other)
Responsible Party: Principal Investigator, Erica Cruvinel, Master degree, PhD student, Federal University of Juiz de Fora
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0022.420.000-11
Record Dates: First submitted 2015-09-24; First posted 2015-10-08 (Estimated); Results first posted 2018-07-30 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2017-10

CONDITIONS: Tobacco Use Cessation; Tobacco Use Disorder
Keywords: Tobacco Use Disorder; Hospitalized patients; Text message; Motivational Interview; Substance-Related Disorders; Behaviors and Mental Disorders
MeSH Terms: conditions — Tobacco Use Cessation; Tobacco Use Disorder; Substance-Related Disorders; Behavior; Mental Disorders | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational Interview plus text message (Experimental): Inside the hospital: All participants have received the written materials. Patients with high tobacco dependence (Fagerstrom screening test score 5 or higher) have received also Nicotine Replacement Therapy (NRT). The written materials provided information on benefits of quitting and strategies for a successful quit plan, including information on relapse prevention. Post discharge extended treatment: Participants in this arm have received a telephone counseling session using a motivational interviewing approach and fifteen or eight days of text messages. The timing, duration, and content of the counseling session were consistent with guideline-based recommendations.
  Interventions: Behavioral: Motivational Interview plus text message
- Control Arm (No Intervention): Inside the hospital: All participants have receive the written materials. Patients with high tobacco dependence (Fagerstrom screening test score 5 or higher) have received also Nicotine Replacement Therapy (NRT). The written materials provided information on benefits of quitting and strategies for a successful quit plan, including information on relapse prevention. Post discharge extended care: None

INTERVENTIONS:
Behavioral: Motivational Interview plus text message — After discharge the experimental group has received extended care including a counseling session and text messages. The session provided basic information about smoking and successful quitting. The counselor has used motivational interview techniques to build coping skills with the goal of helping the participant build and implement a quit plan. The focus was to increase motivation to make quit attempt, including confidence building, medication use, and cessation planning. The session lasted approximately 30 minutes. Participants in the experimental arm were offered up to 30 text messages to help them to implement the quit plan discussed during the phone call. Patients motivated to quit in the next 30 days or those that had already quit have received 30 messages (2 per day) and patients unwilling to quit 16 (2 per day). The messages followed the self efficacy theory.
  Arms: Motivational Interview plus text message

SUMMARY:
This study is a preliminary research aimed to compare the feasibility and effectiveness of motivational interview (MI), Personalized text messages (TM) and usual care for outpatients, with focus on smoking cessation as the main outcome. Smokers patients have received brief interventions and nicotine replacement therapy during the hospitalization. After discharge smokers were allocated into a intervention or control arm. In the first and third months, after randomization, the patients were contact to smoke abstinence assessment.

DETAILED DESCRIPTION:
Background: Research suggests that smokers who receive treatment inside the hospital and post-discharge follow up for at least a month are more likely to quit smoking than those who didn't receive any intervention. The current challenge is to know the best way to support post-discharge quit attempts in the Brazilian context. Objective: The aim of this study was to compare the feasibility and effectiveness of motivational interview (MI) plus Personalized text messages (TM) and usual care for support smoking cessation among post-discharge patients. Methods: All patients admitted to the University Hospital of Juiz de Fora (HU/UFJF), between 06/2015 to 01/2016, were asked about the cigarettes consumption in the last 30 days. Smokers patients received brief interventions and nicotine replacement therapy during the hospitalization. After hospitalization discharge smokers were allocated into a intervention or control arm. The intervention group received a singular MI session by phone and mobile phone TM twice a day during eight or fifteen days. The control group received only usual care available inside the hospital. Results: At the first and third months, after randomization, the patients were contacted for smoke abstinence assessment.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Smoked cigarettes in the last 30 days (even a puff)
* Have own mobile phone
* Have received at least one text message in the last year
* Have no problem with the mobile phone signal

Exclusion Criteria:

* Don't have a mobile phone
* Unstable cognitive or physical condition
* Physical or breath contact restrictions
* Intensive care units

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2015-06; Primary Completion 2016-01 (Actual); Study Completion 2016-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erica Cruvinel, MD, Principal Investigator — Federal University of Juiz de Fora
Locations (1):
- University Federal Hospital of Juiz de Fora, Juiz de Fora, Minas Gerais, Brazil

RESULTS

PARTICIPANT FLOW:
Groups:
- Motivational Interview Plus Text Message: Inside the hospital: All participants will receive the written materials. Patients with high tobacco dependence (Fagerstrom screening test score 5 or higher) will receive also Nicotine replacement therapy. The written materials provide information on, benefits of quitting smoking, and strategies for a successful quit plan, including information on relapse prevention. Post discharge extended treatment: Participants in this arm will receive a telephone counseling session using a motivational interviewing approach and fifteen or eight days of text messages. The timing, duration, and content of the counseling session will be consistent with guideline-based recommendations. Motivational Interview plus text message: After discharge the experimental group will receive extended care including a counseling session and text messages. The session will provide basic information about smoking and successful quitting. The counselor will use motivational interview techniques to build coping
- Control Arm: Inside the hospital: All participants will receive the written materials. Patients with high tobacco dependence (Fagerstrom screening test score 5 or higher) will receive also Nicotine replacement therapy. The written materials provide information on, benefits of quitting smoking and strategies for a successful quit plan, including information on relapse prevention.
  Post discharge extended care: None
Period: Overall Study
Arm/Group | Motivational Interview Plus Text Message | Control Arm
Started | 44 | 22
Completed | 41 | 21
Not Completed | 3 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Unable to reach out post discharge | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Motivational Interview Plus Text Message | Control Arm | Total
Number analyzed (Participants) | 44 | 22 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (12.7) | 48.2 (8.9) | 47.7 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 12 | 32
  Male | 24 | 10 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0
  Race: Asian | 0 | 0 | 0
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race: Black or African American | 6 | 2 | 8
  Race: White | 27 | 17 | 44
  Race: More than one race | 11 | 3 | 14
  Race: Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Self Reported Smoking Abstinence
Description: No smoking (even a puff) in the past 7 days at the first month follow up.
Time Frame: Smoking abstinence at the first month after randomization
Population: The primary analysis was intention-to-treat and involved all patients who were randomly assigned. The 7-day point prevalence abstinence rate was assessed as the first outcome (1-month assessment).
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Interview Plus Text Message | Control Arm
Number analyzed (Participants) | 44 | 22
Participants | 11 | 2
Statistical Analysis 1: Comparison: Motivational Interview Plus Text Message vs Control Arm; Test type: Superiority; Risk Ratio (RR) = 1.35, 95% CI 2-sided [0.99 to 1.85]

2. Secondary Outcome: Daily Cigarettes Consumption at 3 Months Among Continuing Smokers
Description: The experimental group self reported daily cigarettes consumption at the third month after randomization with be compared to the control group.
Time Frame: At the third month after randomization
Population: It was included only patients that were able to be contacted for follow up (per protocol analysis).
Measure: Mean (Standard Deviation); unit: Number of cigarettes smoked per day
Groups:
- Motivational Interview Plus Text Message: Inside the hospital: All participants will receive the written materials. Patients with high tobacco dependence (Fagerstrom screening test score 5 or higher) will receive also Nicotine replacement therapy. The written materials provide information on, benefits of quitting smoking, and strategies for a successful quit plan, including information on relapse prevention. Post discharge extended treatment: Participants in this arm will receive a telephone counseling session using a motivational interviewing approach and fifteen or eight days of text messages. The timing, duration, and content of the counseling session will be consistent with guideline-based recommendations.
  Motivational Interview plus text message: After discharge the experimental group will receive extended care including a counseling session and text messages. The session will provide basic information about smoking and successful quitting. The counselor will use motivational interview techniques to build coping sk
Arm/Group | Motivational Interview Plus Text Message | Control Arm
Number analyzed (Participants) | 41 | 21
Number of cigarettes smoked per day | 12.9 (5.2) | 14.6 (5.5)
Statistical Analysis 1: Comparison: Motivational Interview Plus Text Message vs Control Arm; Test type: Superiority; p = 0.28, t-test, 2 sided

3. Secondary Outcome: Self Reported Seek for Specialized Tobacco Treatment
Description: self reported seek for specialized tobacco treatment after hospitalization
Time Frame: at the third month after randomization
Population: It was included only patients that were able to be contacted for follow up (per protocol analysis).
Measure: Count of Participants; unit: Participants
Groups:
- Motivational Interview Plus Text Message: Inside the hospital: All participants will receive the written materials. Patients with high tobacco dependence (Fagerstrom screening test score 5 or higher) will receive also Nicotine replacement therapy. The written materials provide information on, benefits of quitting smoking, and strategies for a successful quit plan, including information on relapse prevention. Post discharge extended treatment: Participants in this arm will receive a telephone counseling session using a motivational interviewing approach and fifteen or eight days of text messages. The timing, duration, and content of the counseling session will be consistent with guideline-based recommendations.
  Motivational Interview plus text message: After discharge the experimental group will receive extended care including a counseling session and text messages. The session will provide basic information about smoking and successful quitting. The counselor will use motivational interview techniques to build coping s
Arm/Group | Motivational Interview Plus Text Message | Control Arm
Number analyzed (Participants) | 41 | 21
Participants | 0 | 1
Statistical Analysis 1: Comparison: Motivational Interview Plus Text Message vs Control Arm; Test type: Superiority; p = 0.42, Fisher Exact

4. Secondary Outcome: Self Reported Smoking Abstinence
Description: No smoking (even a puff) in the past 7 days at the third month after randomization.
Time Frame: Smoking abstinence at the third month after randomization
Population: The primary analysis was intention-to-treat and involved all patients who were randomly assigned. The 7-day point prevalence abstinence rate, at 3-month assessment, was assessed as a secondary outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Interview Plus Text Message | Control Arm
Number analyzed (Participants) | 44 | 22
Participants | 14 | 2
Statistical Analysis 1: Comparison: Motivational Interview Plus Text Message vs Control Arm; Test type: Superiority; Risk Ratio (RR) = 1.45, 95% CI 2-sided [1.08 to 1.95]

5. Secondary Outcome: Carbon Monoxide Verified Smoking Abstinence
Description: Carbon Monoxide verified Smoking Abstinence at third-month follow up. Abstinence defined as Carbon Monoxide ≤ 6.
Time Frame: At third-month follow up
Population: Intention to Treat Analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Motivational Interview Plus Text Message | Control Arm
Number analyzed (Participants) | 44 | 22
Participants | 9 | 1
Statistical Analysis 1: Comparison: Motivational Interview Plus Text Message vs Control Arm; Test type: Superiority; Risk Ratio (RR) = 1.44, 95% CI 2-sided [1.07 to 1.92]

ADVERSE EVENTS:
Time Frame: Participants received text message during 15 days. Adverse events were not collected during this period.
Groups:
- Motivational Interview Plus Text Message: Inside the hospital: All participants will receive the written materials. Patients with high tobacco dependence (Fagerstrom screening test score 5 or higher) will receive also Nicotine replacement therapy. The written materials provide information on, benefits of quitting smoking, and strategies for a successful quit plan, including information on relapse prevention.
  Post discharge extended treatment: Participants in this arm will receive a telephone counseling session using a motivational interviewing approach and fifteen or eight days of text messages. The timing, duration, and content of the counseling session will be consistent with guideline-based recommendations.Motivational Interview plus text message: After discharge the experimental group will receive extended care including a counseling session and text messages. The session will provide basic information about smoking and successful quitting. The counselor will use motivational interview techniques to build coping
Arm/Group | Motivational Interview Plus Text Message | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No